CLINICAL TRIAL: NCT00747474
Title: A Phase 1 Open-Label, Sequential Dose Escalation Study Investigating the Safety, Tolerability, and Pharmacokinetics of Intravenous Lipotecan® (TLC388 HCl for Injection) When Administered to Patients With Advanced Solid Tumors
Brief Title: Phase I Study of Intravenous Lipotecan® (TLC388 HCl for Injection) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLC388-101
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — TLC 388

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipotecan (Experimental): Intravenous Lipotecan (TLC388 HCl for Injection)
  Interventions: Drug: Lipotecan

INTERVENTIONS:
Drug: Lipotecan — Lipotecan IV day 1, 8, 15
  Other Names: Lipotecan (TLC388)

SUMMARY:
The purpose of this study is to find a safe and tolerable dose of Lipotecan® when administered to patients with advanced solid tumors.

DETAILED DESCRIPTION:
Lipotecan® is a drug product of TLC388 HCl, which is a potent camptothecin analog with cytotoxic activities against a variety of human tumor cell lines in vitro and anti-tumor activities in several xenograft models with human tumor cell lines. Structurally, TLC388 HCl is related to other camptothecins, but it has been chemically modified to improve stability and potency, and to minimize toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients defined by age ≥18 years.
* Pathologically confirmed advanced solid tumors for which standard therapy proven to provide clinical benefit does not exist or is no longer effective
* Evaluable disease, either measurable on imaging or with informative tumor marker(s), by RECIST (Response Evaluation Criteria in Solid Tumors) criteria.

Exclusion Criteria:

* Pregnancy or lactation. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrolment. Male and female patients of childbearing potential must agree to use appropriate birth control (barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine devices) during the entire duration of the study, or the patient must be surgically sterile (with documentation in the patient's medical records).
* Previous malignancy, except for non-basal-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, unless the tumor was treated with curative intent more than 2 years prior to study entry.
* Receipt of more than 3 prior regimens of chemotherapy.
* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to baseline. Receipt of radiotherapy to >25 % of bone marrow. Major surgery within 4 weeks prior to baseline.
* Concomitant treatment with, or anticipated use of, pharmaceutical or herbal agents which are potent inhibitors or inducers of cytochrome P450 enzymes unless approved by the Sponsor.
* Uncontrolled intercurrent illness that would jeopardize patient safety, interfere with the objectives of the protocol, or limit patient compliance with study requirements, as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hsiung Kao, Study Director — Taiwan Liposome Company, Ltd.
Locations (4):
- United States (3):
  - Medical College of Georgia, Augusta, Georgia
  - Bidmc, Dfci, Mgh, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment period was from Sep 2008 to Dec 2010. Patients were recruited from three US clinical sites and one Taiwan site.
Pre-assignment Details: Patients will attend the clinic for a screening visit up to 28 days before receiving, if eligible, the first dose of Lipotecan®.
Groups:
- Cohort 1 (1.5 mg/m^2): Participants received 1.5 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 2 (3 mg/m^2): Participants received 3 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 3 (6 mg/m^2): Participants received 6 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 4 (9 mg/m^2): Participants received 9 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 5 (13.5 mg/m^2): Participants received 13.5 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 6 (20 mg/m^2): Participants received 20 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 7 (30 mg/m^2): Participants received 30 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 8 (40 mg/m^2); Cohort 10 (40 mg/m^2): Participants received 40 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 9 (35 mg/m^2): Participants received 35 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 11 (50 mg/m^2): Participants received 50 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
- Cohort 12 (60 mg/m^2): Participants received 60 mg/m^2/dose, given as a 30 minute IV infusion on Days 1, 8 and 15 of a 28 day cycle. Each 28 day (4 week) period will constitute one cycle of treatment. Dose escalation of Lipotecan® will be based upon the safety and tolerability data from the first treatment cycle in each patient and determined by Safety Review Committee (SRC) for this study.
Period: Cohort 1 (1.5 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2 (3 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3 (6 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4 (9 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 5 (13.5 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 6 (20 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 7 (30 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 8 (40 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — with efficacy and continued treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Cohort 9 (35 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 10 (40 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 11 (50 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 12 (60 mg/m^2) Period
Arm/Group | Cohort 1 (1.5 mg/m^2) | Cohort 2 (3 mg/m^2) | Cohort 3 (6 mg/m^2) | Cohort 4 (9 mg/m^2) | Cohort 5 (13.5 mg/m^2) | Cohort 6 (20 mg/m^2) | Cohort 7 (30 mg/m^2) | Cohort 8 (40 mg/m^2) | Cohort 9 (35 mg/m^2) | Cohort 10 (40 mg/m^2) | Cohort 11 (50 mg/m^2) | Cohort 12 (60 mg/m^2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Population: Lipotecan was administered intravenously on day 1, 8 and 15 of a 28-day cycle.
Arm/Group | Overall Population
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 41
  Taiwan | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Lipotecan
Description: MTD is the highest dose of drug that did not cause an unacceptable side effect (= Dose Limiting Toxicity (DLT)). A 3+3 study design was used to determine MTD. The MTD was the highest dose level at which 0 of 3 or 1 of 6 patients experience a DLT, with the next higher dose having at least 2 of 3 or 2 of 6 patients experiencing a DLT.
Time Frame: First treatment to toxicity up to 42 days
Population: Patients received at least one dose of Lipotecan.
Measure: Number; unit: mg/m^2
Groups:
- All Participants: Lipotecan was administered intravenously on day 1, 8 and 15 of a 28-day cycle according to the dose assigned.
Arm/Group | All Participants
Number analyzed (Participants) | 54
mg/m^2 | 50

2. Secondary Outcome: Anti-tumor Activity
Description: Patients were evaluated by tumor assessment using RECIST guidelines. Possible evaluations include: Complete Response (CR): disappearance of all target lesions. Partial Response (PR): at least a 30% decrease in the size of target lesions. Progressive Disease (PD): at least a 20% increase in the size of target lesions. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From start of treatment assessed every 2 cycles up to 2.5 years
Population: Patients received at least one dose of Lipotecan.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 54
participants
  Complete Response (CR) | 0
  Partitial Response (PR) | 0
  Stable Disease (SD) | 21
  Progression Disease (PD) | 20
  No assessment | 13

3. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with AEs that occurred during treatment and follow-up period (30 days after last treatment). Drug-related AEs and SAEs were followed until resolved or stabilized. AEs were classified by the investigator according to severity graded using CTCAE version 3.0 and relationship to study drug. The severity scale is: Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening or disabling, Grade 5= Death related to AE
Time Frame: an average of 6 months
Population: Patients received at least one dose of Lipotecan
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 54
participants | 54

4. Primary Outcome: Maximum Observed Dose-normalized Plasma Concentration (Cmax) of S,R-TLC388
Description: Drug product Lipotecan consists of TLC388 diastereomers (S,S-TLC388 and S,R-TLC388 in 2:1 ratio). Three metabolites as TLC-U1, TLC-U2 and topotecan were identified in rats, dogs and human.
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
ng/mL | 1.39 (3.21)

5. Primary Outcome: Maximum Observed Dose-normalized Plasma Concentration (Cmax) of S,S-TLC388
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
ng/mL | 2.21 (5.12)

6. Primary Outcome: Maximum Observed Dose-normalized Plasma Concentration (Cmax) of Topotecan
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
ng/mL | 0.82 (0.44)

7. Primary Outcome: Maximum Observed Dose-normalized Plasma Concentration (Cmax) of TLC-U1
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
ng/mL | 5.01 (1.91)

8. Primary Outcome: Maximum Observed Dose-normalized Plasma Concentration (Cmax) of TLC-U2
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1h, 1h30m, 2h, 4h, 8h
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
ng/mL | 1.40 (0.48)

9. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of S,R-TLC388
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 0.47 (0.30)

10. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of S,S-TLC388
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 0.47 (0.30)

11. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Topotecan
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 0.93 (0.82)

12. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of TLC-U1
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 0.45 (0.17)

13. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of TLC-U2
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 0.47 (0.14)

14. Primary Outcome: Dose-normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of S,R-TLC388
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hr*ng/mL | 0.70 (1.63)

15. Primary Outcome: Dose-normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of S,S-TLC388
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hr*ng/mL | 1.04 (2.44)

16. Primary Outcome: Dose-normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of Topotecan
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hr*ng/mL | 3.59 (1.30)

17. Primary Outcome: Dose-normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of TLC-U1
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hr*ng/mL | 7.15 (2.20)

18. Primary Outcome: Dose-normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of TLC-U2
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hr*ng/mL | 2.00 (0.66)

19. Primary Outcome: Plasma Decay Half-Life (t1/2) of S,R-TLC388
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 1.08 (1.77)

20. Primary Outcome: Plasma Decay Half-Life (t1/2) of S,S-TLC388
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 0.75 (1.18)

21. Primary Outcome: Plasma Decay Half-Life (t1/2) of Topotecan
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 6.05 (2.71)

22. Primary Outcome: Plasma Decay Half-Life (t1/2) of TLC-U1
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 3.13 (1.27)

23. Primary Outcome: Plasma Decay Half-Life (t1/2) of TLC-U2
Description: as for outcome 4
Time Frame: 0, 15m, 29m, 33m, 40m, 50m, 1 h, 1h 30m, 2h, 4h, 8h post-dose
Population: Patients complete cycle 1 and 2 treatments without major protocol deviation.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Overall Population
Number analyzed (Participants) | 48
hour | 2.58 (0.62)

ADVERSE EVENTS:
Time Frame: 32 months
Arm/Group | Overall Population
Serious Adverse Events (participants affected / at risk) | 11/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Population (N=54)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 2 (3)
ASTHENIA (General disorders) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2)
CYSTITIS KLEBSIELLA (Infections and infestations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (3)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Population (N=54)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (19)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (7)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (4)
ANAEMIA (Blood and lymphatic system disorders) | 34 (106)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (8)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (4)
CONSTIPATION (Gastrointestinal disorders) | 14 (20)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 (17)
DIARRHOEA (Gastrointestinal disorders) | 15 (25)
DIZZINESS (Nervous system disorders) | 8 (8)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5)
FATIGUE (General disorders) | 22 (48)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 7 (7)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 7 (9)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 7 (7)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOTENSION (Vascular disorders) | 3 (5)
INSOMNIA (Psychiatric disorders) | 5 (5)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 3 (3)
LEUKOPENIA (Blood and lymphatic system disorders) | 13 (23)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (8)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 20 (30)
NEUTROPENIA (Blood and lymphatic system disorders) | 15 (54)
OEDEMA PERIPHERAL (General disorders) | 9 (9)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (8)
PYREXIA (General disorders) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 13 (31)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5)
VOMITING (Gastrointestinal disorders) | 14 (24)
WEIGHT DECREASED (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days